CLINICAL TRIAL: NCT04576156
Title: A Randomized Open-Label, Phase 3 Study to Evaluate Imetelstat (GRN163L) Versus Best Available Therapy (BAT) in Patients With Intermediate-2 or High-risk Myelofibrosis (MF) Relapsed / Refractory (R/R) to Janus Kinase (JAK) Inhibitor
Brief Title: A Study Comparing Imetelstat Versus Best Available Therapy for the Treatment of Intermediate-2 or High-risk Myelofibrosis (MF) Who Have Not Responded to Janus Kinase (JAK)-Inhibitor Treatment
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Geron Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MYF3001; 2020-003288-24 (EudraCT Number); 2023-509120-17-00 (EU CTIS Number)
Record Dates: First submitted 2020-09-18; First posted 2020-10-06 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-10

CONDITIONS: Myelofibrosis
Keywords: Myeloproliferative neoplasms; Polycythemia; Thrombocythemia; Primary myelofibrosis; Janus Kinase-Inhibitor
MeSH Terms: conditions — Primary Myelofibrosis; Myeloproliferative Disorders; Polycythemia; Thrombocytosis | interventions — imetelstat; GRN163L peptide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Imetelstat (Experimental): Participants will receive imetelstat sodium at 9.4 mg/kg intravenous (IV) every 21 days (±3 days), until disease progression or unacceptable toxicity, treatment discontinuation or study end.
  Interventions: Drug: Imetelstat
- Best Available Therapy (BAT) (Active Comparator): Participants will receive BAT (investigator-selected non-JAK-inhibitor treatment), until disease progression or unacceptable toxicity, treatment discontinuation or study end.
  Participants on BAT who meet protocol-defined criteria for progressive disease may crossover to receive imetelstat treatment after sponsor's approval.
  Interventions: Drug: Best Available Therapy (BAT)

INTERVENTIONS:
Drug: Imetelstat — Imetelstat sodium will be given intravenously at 9.4 mg/kg every 21 days, until disease progression or unacceptable toxicity, treatment discontinuation or study end.
  Other Names: GRN163L
  Arms: Imetelstat
Drug: Best Available Therapy (BAT) — Non-JAK-inhibitor treatment will be given, which may include but is not limited to hydroxyurea, thalidomide or an analog of thalidomide, interferon, danazol, hypomethylating agents, chemotherapy or radiotherapy.
  Arms: Best Available Therapy (BAT)

SUMMARY:
The purpose of the study is to evaluate the overall survival of participants treated with imetelstat compared to best available therapy with intermediate-2 or high-risk Myelofibrosis (MF) who are relapsed/refractory (R/R) to Janus Kinase (JAK)-Inhibitor treatment.

DETAILED DESCRIPTION:
This is a multicenter study with 2 arms, and will include 3 phases: a) screening phase of up to 28 days before randomization during which participants will complete a 14-day washout period from all prior therapies including JAK-inhibitor treatment, and the participant's eligibility will be reviewed; b) treatment phase, from randomization until study treatment (imetelstat or BAT) discontinuation; and c) post treatment follow-up phase, that begins when the participant discontinues treatment, and will continue until death, lost to follow-up, withdrawal of consent, or study end, whichever occurs first. Participants will be randomized (2:1) into 2 Arms (Arm A will receive imetelstat and Arm B will receive BAT).

Participants who meet progressive disease criteria and discontinue BAT, may crossover to receive imetelstat treatment after sponsor's approval.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary myelofibrosis according to the revised World Health Organization criteria or post-essential thrombocythemia-MF or post-polycythemia vera-MF according to the IWG-MRT criteria
* Dynamic International Prognostic Scoring System intermediate-2 or high-risk MF
* Relapsed/refractory to JAK-inhibitor treatment as defined in either inclusion (i), (ii) or (iii) and not eligible for allogeneic stem cell transplantation (ASCT) at screening:

  * (i) Treatment with JAK-inhibitor for >= 6 months duration, including at least 2 months at an optimal dose as assessed by the investigator for that participant and at least one of the following:

    1. no decrease in spleen volume (< 10% by MRI or CT) from the start of treatment with JAK-inhibitor
    2. no decrease in spleen size (< 30% by palpation or length by imaging) from the start of treatment with JAK-inhibitor
    3. no decrease in symptoms (< 20% by Myelofibrosis Symptom Assessment Form [MFSAF] or myeloproliferative neoplasm SAF) from the start of treatment with JAK-inhibitor
    4. a score of at least 15 on TSS assessed using the MFSAF v4.0 during screening.
  * (ii) Treatment with JAK-inhibitor treatment for>= 3 months duration with maximal doses (e.g., 20-25 mg twice daily ruxolitinib) for that participant and no decrease in spleen volume/size or symptoms as defined in inclusion criterion (i [a, b, or c]).
  * (iii) Following maximum tolerated doses of JAK inhibitor therapy for ≥3 months duration, having documented relapsed disease defined as either

    1. Increase in spleen volume from time of best response by 25% measured by MRI or CT, or
    2. Increase in spleen size by palpation, CT, or ultrasound

       * (b.i) For splenomegaly of 5-10 cm at the start of JAK inhibitor treatment, at least 100% increase in palpable spleen size from time of best response;
       * (b.ii) For splenomegaly of > 10 cm at the start of JAK inhibitor treatment, at least 50% increase in palpable spleen size from time of best response;

AND not a candidate for further JAK inhibitor at screening per investigator.

* Measurable splenomegaly demonstrated by a palpable spleen measuring >= 5 cm below the left costal margin or a spleen volume >= 450 cm^3 by MRI or CT
* Active symptoms of MF on the MFSAF v4.0 demonstrated by a symptom score of at least 5 points (on a 0 to 10 scale)
* Hematology laboratory test values within the protocol defined limits
* Biochemical laboratory test values must be within protocol defined limits
* Eastern Cooperative Oncology Group Performance Status score of 0, 1, or 2
* Participants should follow protocol defined contraceptives procedures
* A woman of childbearing potential must have a negative serum or urine pregnancy test at screening

Exclusion Criteria:

* Peripheral blood blast count of >= 10% or bone marrow blast count of >=10%
* Known allergies, hypersensitivity, or intolerance to imetelstat or its excipients
* Prior treatment with imetelstat
* Any chemotherapy or MF directed therapy, including investigational drug regardless of class or mechanism of action, immunomodulatory or immunosuppressive therapy, corticosteroids greater than 30 mg/day prednisone or equivalent, and JAK-inhibitor treatment less than equal to 14 days prior to randomization
* Diagnosis or treatment for malignancy other than MF except:

  * Malignancy treated with curative intent and with no known active disease present for >= 3 years before randomization
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated cervical carcinoma in situ without evidence of disease
* Known history of human immunodeficiency virus or any uncontrolled active systemic infection requiring IV antibiotics
* Active systemic hepatitis infection requiring treatment (carriers of hepatitis virus are permitted to enter the study), or any known acute or chronic liver disease requiring treatment unless related to underlying hepatosplenomegaly due to MF
* Major surgery within 28 days prior to randomization
* Any life-threatening illness (e.g., coronavirus disease-2019), medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the participant's safety, interfere with the imetelstat metabolism, or put the study outcomes at undue risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Baseline (Day 1) until End of Study (EOS) (approximately 3 years )]
  Overall survival is defined as the time interval from randomization date to date of death from any cause.

SECONDARY OUTCOMES:
Symptom response rate | Baseline (Day 1), and at Week 24
  The proportion of participants achieving a ≥50% reduction in Total Symptom Score (TSS) measured at Week 24 compared to baseline
Progression-free survival | Baseline (Day 1) until End of Study (EOS) (approximately 3 years)
  Progression-free survival is defined as the time interval from randomization date to the first date of disease progression (worsening splenomegaly or leukemic transformation per 2013 International Working Group - Myeloproliferative Neoplasms Research and Treatment (IWG-MRT) criteria) or death from any cause, whichever occurs first.
Spleen response rate | Baseline (Day 1), and at Week 24
  The proportion of participants who achieve a reduction in spleen volume of ≥ 35% from baseline at Week 24.
Complete remission (CR), partial remission (PR), clinical improvement (CI), spleen response, symptoms response, and anemia response per modified 2013 IWG-MRT criteria | Baseline (Day 1) until End of Treatment (approximately 3 years)
  The proportion of participants achieving CR or PR, CI, spleen response, symptom response, and anemia response per modified 2013 IWG-MRT criteria.
Reduction in the degree of bone marrow fibrosis | Baseline (Day 1) until End of Treatment (approximately 3 years)
  Reduction in the degree of bone marrow fibrosis will be assessed.
Number of Participants with Adverse Events | Screening (Day -28 to -1) until End of Study (approximately 3 years)
  Safety will be assessed based on the incidence and severity (according to the Common Terminology Criteria for Adverse Events) of treatment emergent adverse events from the time of randomization until 30 days after completion of treatment
Assessment of Cmax | Day 1 of all cycles (each cycle is 21 days)
  Maximum Observed Plasma Concentration (Cmax).
Assessment of Tmax | Day 1 of all cycles (each cycle is 21 days)
  Time to reach the maximum observed plasma concentration
Assessment of t1/2 | Day 1 of all cycles (each cycle is 21 days)
  Elimination half-life.
Assessment of AUC | Day 1 of all cycles (each cycle is 21 days)
  Area under the drug concentration-plasma time curve (AUC) from time zero to last measurable concentration
European Organization for Research and Treatment of Cancer Quality-of-Life-Questionnaire-Core-30 (EORTC QLQ-C30) scores | Baseline to End of Study (approximately 3 years)
  Patient-reported outcomes including health-related quality of life, pain, and overall change in participant's health will be assessed using the EORTC QLQ-C30. The EORTC QLQ-C30 includes 30 items resulting in 5 functional scales (physical functioning, role functioning, emotional functioning, cognitive functioning, and social functioning), 1 Global Health Status scale, 3 symptom scales (fatigue, nausea and vomiting, and pain), and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Scores are transformed to a 0 to 100 scale. Higher scores indicated worse outcome.
EuroQol-EQ-5D (EQ-5D-5L) questionnaire scores | Baseline to End of Study (approximately 3 years)
  EQ-5D-5L is a 5 item questionnaire that assesses 5 domains including mobility, self-care, usual activities, pain/discomfort and anxiety/depression plus a visual analog scale rating "health today" with anchors ranging from 0 (worst imaginable health state) to 100 (best imaginable health state).

CONTACTS AND LOCATIONS:
Overall Officials: Faye Feller, Study Director — Geron Corporation
Locations (174):
- United States (18):
  - University of California-San Diego/Moores UCSD Cancer Center, La Jolla, California
  - UCLA David Geffen School of Medicine, Los Angeles, California
  - Smilow Cancer Center at YNHH, New Haven, Connecticut
  - BRCR Medical Center Inc, Plantation, Florida
  - University of South Florida, Tampa, Florida
  - Norton Cancer Institute, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Maryland Oncology Hematology, Rockville, Maryland
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - Prairie Lakes Health Care System, Inc., Watertown, South Dakota
  - Oncology Consultants, Houston, Texas
  - The University of Texas MD, Houston, Texas
  - Community Cancer Trials of Utah, Ogden, Utah
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Hematology Oncology Associates of Fredericksburg, Fredericksburg, Virginia
  - Northwest Medical Specialties PLLC, Seattle, Washington
- Argentina (3):
  - Hospital Aleman, Ciudad de Buenos Aires, Buenos Aires
  - Sanatorio de la Mujer, Rosario, Santa Fe Province
  - Sanatorio Allende, Córdoba
- Australia (4):
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Royal Hobart Hospital, Hobart, Tasmania
  - Epworth Healthcare, Richmond, Victoria
- Austria (4):
  - Krankenhaus Hietzing mit Neurologischem Zentrum Rosenhügel, Wein, Burgenland
  - Krankenhaus der Elisabethinen, Linz, Upper Austria
  - Kepler Universitätsklinikum Gm, Linz, Upper Austria
  - Klinikum Wels-Grieskirchen GmbH, Wels, Upper Austria
- Belgium (5):
  - AZ Klina, Antwerp, Antwerpen
  - UZ Antwerpen, Edegem, Antwerpen
  - Centre Hospitalier de Jolimont, Haine-Saint-Paul, Hainaut
  - Universitair Ziekenhuis Gent, Ghent, Oost-Vlaanderen
  - Universitair Ziekenhuis Brussel - Myeloom Centrum Brussel (MCB), Jette
- Brazil (10):
  - Centro de oncologia Leonardo da Vinci, Fortaleza, Ceará
  - Hospital das Clínicas UFG, Goiânia, Goiás
  - Hospital Erasto Gaertner, Curitiba, Paraná
  - Hospital de Clinicas de Porto Alegre - UFRGS, Porto Alegre, Rio Grande do Sul
  - Centro Gaucho Integrado de Oncologia, Hematologia, Ensino e Pesquisa LTDA, Porto Alegre, Rio Grande do Sul
  - Instituto de Educação, Pesquisa e Gestão em Saúde, São Paulo, São Paulo
  - Hospital Israelita Albert Einstein, São Paulo, São Paulo
  - Fundacao Doutor Amaral Carvalho / Hospital Amaral Carvalho, São Paulo, São Paulo
  - CEPON Centro de Pesquisas Oncologicas SC, Florianópolis
  - Hospital A.C.Camargo Cancer Center - Clinical Oncology, São Paulo
- Bulgaria (2):
  - UMBAL Sveti Georgi, Plovdiv, Plovdiv
  - Specialized Hospital for Active Therapy of Hematological dis, Sofia, Sofia
- Colombia (3):
  - Oncologos del Occidente S.A, Pereira, Risaralda Department
  - Hospital Pablo Tobon Uribe, Antioquia
  - Centro Medico Imbanaco de Cali S.A., Cali
- Odense University Hospital - Hematology, Odense, Denmark
- France (10):
  - Centre Hospitalier Lyon, Pierre-Bénite, Auvergne-Rhône-Alpes
  - CHU Bretonneau, Tours, Indre-et-Loire
  - Hopital Bicetre, Paris, Le Kremlin-Bicêtre
  - CHU De Nantes - Hematologie, Nantes, Loire-Atlantique
  - CHU de Nice - Hopital de l'Archet II - Pharmacie, Nice, Nice Cedex 3
  - Hospital CENTRE HOSPITALIER AVIGNON, Avignon, Provence-Alpes-Côte d'Azur Region
  - Centre Hospitalier Du Mans - Cancérologie Médicale, Le Mans, Sarthe
  - CHRU Brest - Hôpital Morvan, Brest
  - CHU - HÃ´pital Saint Louis - Centre D'Investigations Cliniq, Paris
  - Hopital Cochin - Aphp Hôpitaux Universitaires Paris Centre, Paris, Île-de-France Region
- Georgia (5):
  - J.S.C."K.Eristavi National Cen, Tbilisi, K'alak'i T'bilisi
  - Ltd "Medinvest - Institute of Hematology and Trans, Tbilisi, K'alak'i T'bilisi
  - LTD Israeli-Georgian Medical R, Tbilisi
  - M.Zodelava Hematology Center L, Tbilisi
  - Multi Profile Clinic Consilium, Tbilisi
- Germany (6):
  - Universitätsklinikum Mannheim - University of Heidelberg, Mannheim, Baden-Wurttemberg
  - Universitätsklinikum Tübingen, Tübingen, Baden-Wurttemberg
  - Universitätsklinikum Carl Gust, Dresden, Hamburg
  - Klinikum Kempten-Oberallgaeu GmbH, Kempten, Rhineland-Palatinate
  - Universitätsklinikum Leipzig AöR, Leipzig, Saxony
  - Martin-Luther-Universität Halle-Wittenberg, Halle, Saxony-Anhalt
- Szabolcs-Szatmár-Bereg Megyei Önkormányzat Jósa András, Nyíregyháza, Hungary
- India (11):
  - Nirmal Hospital - Hematology, Surat, Gujarat
  - St. John's Medical College Hospital, Bangalore, Karnataka
  - Fortis Hospital 154/9, Bengaluru, Karnataka
  - All India Institute of Medical Sciences, Dept. of Hematology, New Delhi (All India Institute Of Medical Sciences), New Delhi, National Capital Territory of Delhi
  - Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi
  - Fortis Memorial Research Institute, Gūrgaon, New Delhi
  - All India Institute of Medical Sciences, Bhubaneswar, Odisha
  - Nilratan Sircar Medical College, Kolkata, West Bengal
  - Narayana Hrudayalaya Hospital, Hyderabad
  - Deenanath Mangeshkar Hospital & Research Center, Pune
  - Sahyadri Specialty Hospital, Pune
- Israel (9):
  - Kaplan Medical Center, Rehovot, Central District
  - Shamir Medical Center (Assaf Harofeh), Ẕerifin, Central District
  - Hadassah Medical Organization, Jerusalem, Jerusalem
  - Western Galilee Hospital - Nahariya, Nahariya, Northern District
  - Assuta Ashdod University Hospi, Ashdod, Southern District
  - Barzilai Medical Center, Ashkelon, Southern District
  - Soroka Medical Center - Hematology Institute, Beersheba
  - Bnai Zion Medical Center, Haifa
  - Carmel MC, Haifa
- Italy (23):
  - PO Civile SS.Antonio e Biagio, Alessandria, Alessandria
  - A.O.di Bologna Policl.S.Orsola, Bologna, Bologna
  - Arcispedale S.Anna - Ematologi, Cona, Ferrara
  - AOU Careggi, Florence, Firenze
  - IRCCS Ospedale Policlinico San Martino, Genova, Genova
  - Clinica Ematologica, Univ. Deg, Genova, Genova
  - Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico, Milan, Milano
  - Ospedale Civile S.Maria delle Croci, AUSL Ravenna, Ravenna, Ravenna
  - Arcispedale S Maria Nuova, AO di Reggio Emilia, Reggio Calabria, Reggio Calabria
  - Azienda Ospedaliera Bianchi-Me, Reggio Calabria, Reggio Calabria
  - AUSL di Rimini Ospedale Infermi di Rimini, Rimini, Rimini
  - Policlinico Universitario Agostino Gemelli, Roma, Roma
  - AOU San Luigi Gonzaga, Orbassano, Torino
  - AOU Città della Salute e della Scienza di Torino, Torino, Torino
  - Ospedale di Circolo, PO Varese, Varese, Varese
  - Ospedale S.Bortolo, AULSS n.6, Vicenza, Vicenza
  - Presidio Ospedaliero Garibaldi, Catania
  - Irccs Irst, Meldola
  - Ospedale San Raffaele, Milan
  - ASST Grande Ospedale Metropoli, Milan
  - Azienda Ospedaliera San Gerard, Monza
  - AOU Federico II, Napoli
  - ASL Roma 2 - PO "S. Eugenio", Roma
- Malaysia (5):
  - Hospital Pulau Pinang, Pulau Pinang, Georgetown
  - Hospital Sultanah Aminah Johor Bahru, Johor Bahru, Johor
  - Hospital Raja Perempuan Zainab II, Kota Bharu, Kelantan
  - Sarawak General Hospital, Kuching, Sarawak
  - Hospital Ampang, Ampang, Selangor
- Poland (4):
  - Ars Medical Sp. z o.o., Piła, Greater Poland Voivodeship
  - Centrum Medyczne Pratia Poznan, Skórzewo, Greater Poland Voivodeship
  - Pratia Onkologia Katowice, Katowice, Silesian Voivodeship
  - Wojewodzki Szpital Specjalistyczny, Biała Podlaska
- Portugal (4):
  - CCA-Braga. Centro Clínico Académico - Hospital Braga, Braga, Braga District
  - Centro Clinico Fundacao Champalimaud, Lisbon, Lisbon District
  - H. Santa Maria. Centro Hospita, Lisbon, Lisbon District
  - H. São Francisco Xavier-Centro, Lisbon
- Russia (4):
  - MONIKI - Oncology, Moscow, Moscow Oblast
  - MUZ City Clinical Hospital # 2, Novosibirsk, Novosibirsk Oblast
  - Budgetary Healthcare Institution of Omsk Region, Omsk
  - GOU VPO Saratov State Medical University n.a. V.I., Saratov
- Singapore (2):
  - National University Cancer Institute (NCIS), Singapore, Central Singapore
  - Singapore General Hospital, Singapore, Central Singapore
- South Korea (12):
  - Inje University Busan Paik Hos, Busan, Busan Gwang'Yeogsi [Pusan-Kwangyokshi]
  - Inje University Haeundae Paik Hospital, Busan, Busan Gwang'Yeogsi [Pusan-Kwangyokshi]
  - National Cancer Institute Center for Cancer Research, Goyang-si, Gyeonggido
  - Gachon University Gil Medical Center, Incheon, Incheon Gwang'Yeogsi [Inch'n-Kwangyokshi]
  - Korea University Anam Hospital, Seoul, Seoul Teugbyeolsi [Seoul-T'Ukpyolshi]
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul, Seoul Teugbyeolsi [Seoul-T'Ukpyolshi]
  - Korea University Guro Hospital, Seoul, Seoul Teugbyeolsi [Seoul-T'Ukpyolshi]
  - Samsung Medical Center, Seoul, Seoul Teugbyeolsi [Seoul-T'Ukpyolshi]
  - Seoul National University Hospital - Department of Internal, Seoul, Seoul Teugbyeolsi [Seoul-T'Ukp
  - Pusan National University Hospital - Hematology and Oncology, Busan
  - The Catholic University of Korea, Seongdong
  - Severance Hospital, Yonsei Uni, Seoul
- Spain (14):
  - H.G.U. Alicante, Alicante, Alicante
  - Institut Català d'Oncologia-Ho, Badalona, Barcelona
  - C.S. Parc Tauli, Sabadell, Barcelona
  - Hospital Universitario de Gran, Las Palmas de Gran Canaria, Canary Islands
  - H. San Pedro de Alcántara, Cáceres, Cáceres
  - ICO-Hospital Universitari de G, Girona, Girona
  - Hospital Universitario Virgen, Granada, Granada
  - Hospital U. 12 Octubre, Madrid, Madrid
  - H.U. La Paz, Madrid, Madrid
  - H.U.V. de la Victoria, Málaga, Málaga
  - H.U. Ribera de Alzira, Alzira, Valencia
  - H. Quirón Zaragoza, Zaragoza, Zaragoza
  - Hospital Universitario Fundaci, Madrid
  - Hospital Universitario de Salamanco, Salamanca
- Taiwan (3):
  - Chang Gung Medical Foundation, Chiayi City, Chiayi
  - Tri-Service General Hospital, Taipei, Taipei
  - China Medical University Hospital - Hematology/Onc, Taichung
- Turkey (Türkiye) (8):
  - Ankara University Medical Facu, Ankara, Ankara
  - Istanbul üniversitesi cerrahpaşa, Istanbul, Istanbul
  - Medipol Bagcilar Mega Hospital, Istanbul, Istanbul
  - Marmara university pendik training and research hospital, Istanbul, Istanbul
  - Ege Universitesi Tip Fakultesi, Izmir, İzmir
  - Medical Park Mersin Hastanesi, Mersin, Mersin
  - Sakarya Research and Training Hospital - Medical Oncology, Adapazarı
  - Gazi University Medical Faculty, Ankara
- United Kingdom (3):
  - St Bartholomew's Hospital, London
  - Guys and St Thomas' Hospital, London
  - Oxford University Hospitals, Oxford

REFERENCES:
- [Derived] Mascarenhas J, Harrison CN, Kiladjian JJ, Komrokji RS, Koschmieder S, Vannucchi AM, Berry T, Redding D, Sherman L, Dougherty S, Peng L, Sun L, Huang F, Wan Y, Feller FM, Rizo A, Verstovsek S. Imetelstat in intermediate-2 or high-risk myelofibrosis refractory to JAK inhibitor: IMpactMF phase III study design. Future Oncol. 2022 Jul;18(22):2393-2402. doi: 10.2217/fon-2022-0235. Epub 2022 May 5. PMID 35510486